CLINICAL TRIAL: NCT04088708
Title: Role of Gut Microbe Composition in Psychosocial Symptom Response to Exercise Training in Breast Cancer Survivors (ROME Study)
Brief Title: Gut Microbe Composition, Exercise, and Breast Breast Cancer Survivors
Acronym: ROME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura Q. Rogers, MD, MPH, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-30000320; R01CA235598 (NIH)
Record Dates: First submitted 2019-08-03; First posted 2019-09-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Gut Microbiome; Exercise; Fatigue
Keywords: breast cancer; fatigue; exercise; psychosocial outcomes; inflammation; gut microbiome
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Fatigue; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to participant study group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise Training (Experimental): Progressive aerobic exercise training sessions supervised by exercise specialists who have experience training cancer survivors.
  Interventions: Other: Aerobic Exercise Training
- Attention Control (Active Comparator): The non-aerobic exercise attention control condition will control for the effects of attention with flexibility/toning activities.
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Aerobic Exercise Training — Each session will last 20 to 60 minutes depending on the stage of progression (shorter duration in the first few weeks). Sessions will occur on nonconsecutive days of the week. Moderate-intensity, continuous aerobic exercise will be used to target large muscle groups (e.g., legs) with the principal goal of increasing cardiorespiratory fitness. Exercise intensity will be gradually increased. To mitigate stagnation and support continued improvement of cardiorespiratory fitness, high-intensity interval exercise will be added in later weeks of the intervention.
  Arms: Aerobic Exercise Training
Other: Attention Control — The flexibility/toning control condition will be delivered using the same frequency as the aerobic condition (i.e., 3 times per week) and use light resistance bands of least difficulty. The flexibility/toning sessions will last about 40 minutes, be led by trained exercise specialists. Flexibility/toning activities will target the head/neck, shoulder, elbow/forearm, hand/wrist, trunk/hip, and ankle/foot. The progression of activities over the 10-week period will involve performing additional exercises and sets along with using progressively thicker elastic resistance bands (i.e., Thera-bands) that provide minimal resistance.
  Arms: Attention Control

SUMMARY:
The primary goal of this project is to determine the effects of exercise on the gut microbiome in breast cancer survivors and determine how these changes may relate to psychosocial symptoms such as fatigue.

DETAILED DESCRIPTION:
Cancer survivors are at increased risk of gut bacteria communities that can negatively impact health and energy level and it is possible that exercise can cause healthy changes in these communities. Through careful design, this study will use a controlled-feeding diet and 10 weeks of exercise training to determine exercise effects on the number, distribution, and types of bacteria in the gut of breast cancer survivors. These changes will then be linked to fatigue and physiologic effects of exercise to determine how the information can be used to enhance exercise benefits and identify new treatment strategies leveraging changes in gut bacteria communities.

ELIGIBILITY:
Inclusion criteria:

* Women ages 18 to 74 years with a history of breast cancer stage 0, I, II, or III,
* ≥ 1-year post-completion of primary treatment for breast cancer (chemotherapy and/or radiation),
* Average fatigue over the past week rated as ≥3 on a 1 to 10 Likert scale, cut point chosen because it is a clinically meaningful cutpoint,93
* English speaking,
* Physician medical clearance for study participation,
* Able to ambulate without assistance,
* No antibiotics for the past 90 days,
* Willing to avoid taking probiotics for the duration of the study
* Peak VO2 <30 ml/kg/min (note: will measure peak VO2 if the participant meets all other criteria and consents to lab-based screening).

Exclusion criteria:

* Metastatic or recurrent cancer
* Another diagnosis of cancer in the past 5 years (not including skin or cervical cancer in situ), 3)
* Unstable angina
* New York Heart Association class II, III, or IV congestive heart failure
* Uncontrolled asthma
* Interstitial lung disease
* Current steroid use
* Having been told by a physician to only do exercise prescribed by a physician
* Dementia or organic brain syndrome
* Schizophrenia or active psychosis
* Connective tissue or rheumatologic disease (i.e., systemic lupus erythematosus, rheumatoid arthritis, amyloidosis, Reiter's syndrome, psoriatic arthritis, mixed connective tissue disease, Sjögren's syndrome, CREST syndrome, polymyositis, dermatomyositis, progressive systemic sclerosis, vasculitis, polymyalgia rheumatic, temporal arteritis)
* Anticipate elective surgery during the study period
* Anticipate changes in usual medications during the study period
* Plan to move residence out of the local area during the study period
* Plan to travel out of the local area for >1 week during study participation
* Contraindication to engaging in moderate-to-vigorous intensity aerobic exercise
* Currently pregnant or anticipate pregnancy during study participation
* Live or work >50 miles from study site or do not have transportation to study site
* BMI >50
* Anticipate needing antibiotics during the study period

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation
Enrollment: 126 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Composition of gut microbiota as measured by fecal samples | Baseline
  Using standard diversity and taxa comparison metrics
Composition of gut microbiota as measured by fecal samples | 5 weeks after baseline
  Using standard diversity and taxa comparison metrics
Composition of gut microbiota as measured by fecal samples | 10 weeks after baseline
  Using standard diversity and taxa comparison metrics
Composition of gut microbiota as measured by fecal samples | 15 weeks after baseline
  Using standard diversity and taxa comparison metrics

SECONDARY OUTCOMES:
Systemic inflammation tested via blood biomarkers | Baseline
  Blood samples will be analyzed for markers of inflammation (IL-6, IL-10)
Systemic inflammation tested via blood biomarkers | 5 weeks after baseline
  Blood samples will be analyzed for markers of inflammation (IL-6, IL-10)
Systemic inflammation tested via biomarkers | 10 weeks after baseline
  Blood samples will be analyzed for markers of inflammation (IL-6, IL-10)
Systemic inflammation tested via blood biomarkers | 15 weeks after baseline
  Blood samples will be analyzed for markers of inflammation (IL-6, IL-10)
Autonomic nervous system measured through non-invasive ECG | Baseline
  Using a Actiheart 5 to measure heart rate variability and impedance cardiography while resting quietly
Autonomic nervous system measured through non-invasive ECG | 5 weeks after baseline
  Using a Actiheart 5 to measure heart rate variability and impedance cardiography while resting quietly
Autonomic nervous system measured through non-invasive ECG | 10 weeks after baseline
  Using a Actiheart 5 to measure heart rate variability and impedance cardiography while resting quietly
Autonomic nervous system measured through non-invasive ECG | 15 weeks after baseline
  Using a Actiheart 5 to measure heart rate variability and impedance cardiography while resting quietly
Concentration of cortisol measured through hair sample | Baseline
  Hormone change that is associated with stress
Concentration of cortisol measured through hair sample | 5 weeks after baseline
  Hormone change that is associated with stress
Concentration of cortisol measured through hair sample | 10 weeks after baseline
  Hormone change that is associated with stress
Concentration of cortisol measured through hair sample | 15 weeks after baseline
  Hormone change that is associated with stress
Fatigue measured through fatigue specific questionnaire | Baseline
  Fatigue Symptom Inventory which contains 13 items (fatigue intensity = mean of 4 items, 1 to 10 scale; fatigue interference = mean of 7 items, 0 to 10 scale; 2 general fatigue items = 0 to 7 scale and 1 to 10 scale); higher score indicates greater fatigue
Fatigue measured through fatigue specific questionnaire | 5 weeks after baseline
  Fatigue Symptom Inventory which contains 13 items (fatigue intensity = mean of 4 items, 1 to 10 scale; fatigue interference = mean of 7 items, 0 to 10 scale; 2 general fatigue items = 0 to 7 scale and 1 to 10 scale); higher score indicates greater fatigue
Fatigue measured through fatigue specific questionnaire | 10 weeks after baseline
  Fatigue Symptom Inventory which contains 13 items (fatigue intensity = mean of 4 items, 1 to 10 scale; fatigue interference = mean of 7 items, 0 to 10 scale; 2 general fatigue items = 0 to 7 scale and 1 to 10 scale); higher score indicates greater fatigue
Fatigue measured through fatigue specific questionnaire | 15 weeks after baseline
  Fatigue Symptom Inventory which contains 13 items (fatigue intensity = mean of 4 items, 1 to 10 scale; fatigue interference = mean of 7 items, 0 to 10 scale; 2 general fatigue items = 0 to 7 scale and 1 to 10 scale); higher score indicates greater fatigue

OTHER OUTCOMES:
Peak VO2 (oxygen consumption) measured via modified Balke treadmill protocol | Baseline
  Cardiorespiratory fitness test on a treadmill
Peak VO2 (oxygen consumption) measured via modified Balke treadmill protocol | 5 weeks after baseline
  Cardiorespiratory fitness test on a treadmill
Peak VO2 (oxygen consumption) measured via modified Balke treadmill protocol | 10 weeks after baseline
  Cardiorespiratory fitness test on a treadmill
Peak VO2 (oxygen consumption) measured via modified Balke treadmill protocol | 15 weeks after baseline
  Cardiorespiratory fitness test on a treadmill
Walking Economy measured via 6 minute treadmill test | Baseline
  Fitness test on a treadmill
Walking Economy measured via 6 minute treadmill test | 5 weeks after baseline
  Fitness test on a treadmill
Walking Economy measured via 6 minute treadmill test | 10 weeks after baseline
  Fitness test on a treadmill
Walking Economy measured via 6 minute treadmill test | 15 weeks after baseline
  Fitness test on a treadmill
Accelerometer Measured Free-living physical activity (e.g., minutes of activity) | Baseline
  Motion sensor measures physical activity not observed during intervention activities
Accelerometer Measured Free-living physical activity (e.g., minutes of activity) | 5 weeks after baseline
  Motion sensor measures physical activity not observed during intervention activities
Accelerometer Measured Free-living physical activity (e.g., minutes of activity) | 10 weeks after baseline
  Motion sensor measures physical activity not observed during intervention activities
Accelerometer Measured Free-living physical activity (e.g., minutes of activity) | 15 weeks after baseline
  Motion sensor measures physical activity not observed during intervention activities
Body composition using a dual energy x-ray absorptiometry | Baseline
  Measurement of body composition
Body composition using a dual energy x-ray absorptiometry | 5 weeks after baseline
  Measurement of body composition
Body composition using a dual energy x-ray absorptiometry | 10 weeks after baseline
  Measurement of body composition
Body composition using a dual energy x-ray absorptiometry | 15 weeks after baseline
  Measurement of body composition
FACT-B self-administered survey measuring quality of life | Baseline
  Functional Assessment of Cancer Therapy (FACT) - Breast quality of life scale (37 items; 0 to 4 scale; range is 0 to 148); higher score indicates better quality of life
FACT-B self-administered survey measuring quality of life | 5 weeks after baseline
  Functional Assessment of Cancer Therapy (FACT) - Breast quality of life scale (37 items; 0 to 4 scale; range is 0 to 148); higher score indicates better quality of life
FACT-B self-administered survey measuring quality of life | 10 weeks after baseline
  Functional Assessment of Cancer Therapy (FACT) - Breast quality of life scale (37 items; 0 to 4 scale; range is 0 to 148); higher score indicates better quality of life
FACT-B self-administered survey measuring quality of life | 15 weeks after baseline
  Functional Assessment of Cancer Therapy (FACT) - Breast quality of life scale (37 items; 0 to 4 scale; range is 0 to 148); higher score indicates better quality of life
Self-efficacy by self-administered survey | Baseline
  Self-efficacy measured with 15 items (barriers self-efficacy = 9 items and walking self-efficacy = 6 items, mean of 0% to 100% Scale, range is 0% to 100%); higher score indicates higher self-efficacy.
Self-efficacy by self-administered survey | 6 weeks after baseline
  Self-efficacy measured with 15 items (barriers self-efficacy = 9 items and walking self-efficacy = 6 items, mean of 0% to 100% Scale, range is 0% to 100%); higher score indicates higher self-efficacy.
Self-efficacy by self-administered survey | 10 weeks after baseline
  Self-efficacy measured with 15 items (barriers self-efficacy = 9 items and walking self-efficacy = 6 items, mean of 0% to 100% Scale, range is 0% to 100%); higher score indicates higher self-efficacy.
Self-efficacy by self-administered survey | 15 weeks after baseline
  Self-efficacy measured with 15 items (barriers self-efficacy = 9 items and walking self-efficacy = 6 items, mean of 0% to 100% Scale, range is 0% to 100%); higher score indicates higher self-efficacy.
Self-administered survey measuring mood and stress | Baseline
  Measurement of mood and stress after a traumatic experience, Civilian PTSD ( total of 17 items, 1 to 5 scale; range of 17 to 85) higher scores indicate greater PTSD. Perceived Stress Scale - 10 (10 items, 1 to 5 scale; 10 to 50 range) higher score indicates greater perceived stress.
Self-administered survey measuring mood and stress | 5 weeks after baseline
  Measurement of mood and stress after a traumatic experience, Civilian PTSD ( total of 17 items, 1 to 5 scale; range of 17 to 85) higher scores indicate greater PTSD. Perceived Stress Scale - 10 (10 items, 1 to 5 scale; 10 to 50 range) higher score indicates greater perceived stress.
Self-administered survey measuring mood and stress | 10 weeks after baseline
  Measurement of mood and stress after a traumatic experience, Civilian PTSD ( total of 17 items, 1 to 5 scale; range of 17 to 85) higher scores indicate greater PTSD. Perceived Stress Scale - 10 (10 items, 1 to 5 scale; 10 to 50 range) higher score indicates greater perceived stress.
Self-administered survey measuring mood and stress | 15 weeks after baseline
  Measurement of mood and stress after a traumatic experience, Civilian PTSD ( total of 17 items, 1 to 5 scale; range of 17 to 85) higher scores indicate greater PTSD. Perceived Stress Scale - 10 (10 items, 1 to 5 scale; 10 to 50 range) higher score indicates greater perceived stress.
Self-administered survey measuring memory | Baseline
  Measurement of memory through frequency of forgetting scale (total of 10 items, 1 to 7 scale; range of 10 to 70) higher score indicate lower frequency of forgetting and higher level of memory.
Self-administered survey measuring memory | 5 weeks after baseline
  Measurement of memory through frequency of forgetting scale (total of 10 items, 1 to 7 scale; range of 10 to 70) higher score indicate lower frequency of forgetting and higher level of memory.
Self-administered survey measuring memory | 10 weeks after baseline
  Measurement of memory through frequency of forgetting scale (total of 10 items, 1 to 7 scale; range of 10 to 70) higher score indicate lower frequency of forgetting and higher level of memory.
Self-administered survey measuring memory | 15 weeks after baseline
  Measurement of memory through frequency of forgetting scale (total of 10 items, 1 to 7 scale; range of 10 to 70) higher score indicate lower frequency of forgetting and higher level of memory.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Q Rogers, MD, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data collected with National Institutes of Health (NIH) funding and made public through publication in a peer-reviewed format will thereafter be available on request to faculty of institutions with Public Health Service (PHS) assurance. For sharing data and specimens from individual human subjects, the investigators will comply with all relevant policies including the "Standards for Privacy of Individually Identifiable Health Information" rule of the Health Insurance Portability and Accountability Act (HIPAA). For sharing data, the investigators will comply with the requirements of the Final NIH Statement on Sharing Research Data (NOT-OD-03-032), the Policy for Sharing of Data Obtained in NIH Supported or Conducted Genome-Wide Association Studies (GWAS) (NOT-OD-07-088), the NIH Genomic Data Sharing Policy (NOT-OD-14-124), and all other existing, updated, and new requirements as stated by NIH policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: To be determined
Access Criteria: To be determined

REFERENCES:
- [Derived] Little RB, Carter SJ, Motl RW, Hunter G, Cook A, Liu N, Krontiras H, Lefkowitz EJ, Turan B, Schleicher E, Rogers LQ. Role of Gut Microbe Composition in Psychosocial Symptom Response to Exercise Training in Breast Cancer Survivors (ROME) study: protocol for a randomised controlled trial. BMJ Open. 2024 May 3;14(5):e081660. doi: 10.1136/bmjopen-2023-081660. PMID 38702085